CLINICAL TRIAL: NCT01194531
Title: IPSO Trial - Impact of Parental Support on Pregnancy Outcomes: A Multi-Center, Randomized, Open-Label Study to Evaluate the Implantation and Pregnancy Rates Following 24 Chromosome Aneuploidy Screening With Parental Support in Patients Undergoing In Vitro Fertilization (IVF)
Brief Title: Impact of Parental Support on Pregnancy Outcomes (IPSO) Trial- Day 3 Preimplantation Genetic Screening (PGS) With Day 5 Fresh Transfer
Acronym: IPSO
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Slow enrollment and Natera is transitioning to a new PGS testing platform.
Sponsor: Natera, Inc. (Industry)
Collaborators: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: IVF006-D3
Record Dates: First submitted 2010-08-02; First posted 2010-09-03 (Estimated); Results first posted 2014-11-13 (Estimated); Last update posted 2014-11-25 (Estimated); Status verified 2014-11

CONDITIONS: Preimplantation Gentic Screening (PGS); In Vitro Fertilization (IVF); Preimplantation Genetic Diagnosis (PGD)
Keywords: Preimplantation Gentic Screening; PGS; In Vitro Fertilization; IVF; Preimplantation Genetic Diagnosis; PGD
MeSH Terms: interventions — Preimplantation Diagnosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CONTROL arm (No Intervention): Subjects assigned to this arm of the study will receive no PGS testing.
- TEST arm (Other): Subjects assigned to this arm of the study will receive PGS testing.
  Interventions: Device: 24 Chromosome Aneuploidy Screening with Parental Support

INTERVENTIONS:
Device: 24 Chromosome Aneuploidy Screening with Parental Support — Preimplantation Genetic Screening (PGS)
  Other Names: Preimplantation Genetic Diagnosis (PGD)
  Arms: TEST arm

SUMMARY:
Natera is recruiting patients for a research study evaluating pregnancy and implantation rates in women undergoing In Vitro Fertilization (IVF) and Preimplantation Genetic Screening (PGS). PGS is also referred to as Preimplantation Genetic Diagnosis (PGD) for aneuploidy.

Healthy women undergoing IVF who are between the ages of 35 to 42 years are being recruited to participate in a randomized study.

The purpose of this study is to determine whether PGS- testing of embryos created during IVF for chromosomal abnormalities, prior to transfer to the uterus- improves pregnancy and implantation rates in patients when compared to patients whose embryos are not tested. PGS will be conducted using 24 Chromosome Aneuploidy Screening with Parental Support from Natera.

All subjects who qualify and enroll will receive discounted IVF medications (both TEST and CONTROL arms). If you become pregnant during the study, you will receive a small payment for providing information about your pregnancy and birth. If you are assigned to the TEST arm of the study you will receive free PGS.

DETAILED DESCRIPTION:
If you meet the criteria below, you may be a candidate for this study. To participate in the study you must:

* Be a healthy, pre-menopausal female, 35-42 years of age
* Have a history of less than 3 consecutive miscarriages and no more than one failed IVF cycle
* Agree to use Ferring Pharmaceutical products during stimulation
* Agree to be randomly assigned to either the arm of the study receiving PGS (TEST arm)or the arm receiving no additional testing (CONTROL arm)

Additional screening will be conducted to determine if you are eligible to enroll.

All subjects who qualify and enroll will receive discounted IVF medications. If you become pregnant during the study, you will receive a small payment for providing information about your pregnancy and birth. If you are assigned to the TEST arm of the study you will receive free PGS.

ELIGIBILITY:
Inclusion Criteria:

* Must agree to a follow-up visit at approximately 4-8 weeks gestation and a follow up phone call at 20 and 40 weeks gestation/livebirth. For patients assigned to the TEST group must agree to PGD testing and collection of buccal swab sample on newborn
* At least 10 eggs retrieved
* Must agree to use only Ferring products during stimulation
* Normal uterine cavity detected on hysterosalpingogram (HSG), saline infusion sonogram (SIS), or hysteroscopy
* Signed consent form

Exclusion Criteria:

* FSH ≥10 IU/L within past year prior to screening
* 2 or more previously failed IVF cycles
* Gestational or surrogate carrier, donor oocyte, donor sperm
* History of recurrent pregnancy loss (3 or more consecutive miscarriages)
* Severe male factor infertility defined as ejaculate sperm of < 1million sperm/ml, or sperm obtained through testicular biopsy
* Gender selection as primary indication
* Maternal disease that is not clinically stable and known to impact the ability to become pregnant or carry a pregnancy to term (lupus, chronic liver or kidney disease, body mass index (BMI) >35, uncontrolled hypertension, anti-phospholipid antibody, thrombophilia, insulin dependent diabetes)
* Refusal or inability to comply with the requirements of the Protocol for any reason, including scheduled clinic visits and laboratory tests
* Participation in any experimental drug study within 30 days prior to Screening
* Prior hypersensitivity to any of the protocol drugs
* Known history conveying increased risk for chromosome abnormality (beyond maternal age) or genetic disease in offspring

Ages: 35 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2010-09; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Huntington Reproductive Center, Laguna Hills, California
  - Shady Grove Fertility RSC, Washington D.C., District of Columbia
  - Florida Fertility Institute/ Women's Medical Research Group, LLC, Clearwater, Florida
  - Atlanta Center for Reproductive Medicine, Atlanta, Georgia
  - Fertility Centers of Illinois, Chicago, Illinois
  - Boston IVF, Boston, Massachusetts
  - The Nevada Center for Reproductive Medicine, Reno, Nevada
  - Main Line Fertility, Bryn Mawr, Pennsylvania
  - Fertility Specialist of Houston, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CONTROL Arm | TEST Arm
Started | 29 | 30
Completed | 24 | 27
Not Completed | 5 | 3
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Protocol Violation | 4 | 1
Not completed — Physician Decision | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CONTROL Arm | TEST Arm | Total
Number analyzed (Participants) | 29 | 30 | 59
Age, Continuous [Mean (Full Range); unit: years] | 38 [35 to 41] | 37.3 [35 to 42] | 37.7 [35 to 42]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 30 | 59
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Implantation Rate
Description: Implantation rate is defined as the ratio between the number of gestational sacs with a fetal heartbeat and the total number of embryos transferred.
Time Frame: Data is collected at approximately 4-6 weeks gestation, 20 weeks gestation and 40 weeks gestation.
Population: Patients who reached embryo transfer were included in this analysis.
Measure: Number; unit: percentage of implantation per group
Arm/Group | CONTROL Arm | TEST Arm
Number analyzed (Participants) | 22 | 21
percentage of implantation per group | 24 | 35

ADVERSE EVENTS:
Arm/Group | CONTROL Arm | TEST Arm
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/30
Other Adverse Events (participants affected / at risk) | 0/29 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Each PI signed an agreement that all data, analyses, information and materials prepared or derived as a direct result of the Study are required to be provided to the sponsor and in accordance with the Protocol, whether preliminary or final (the "Study Results") shall be property of the sponsor. Site may utilize the Study Results for patient care and for it's own internal education purposes.